CLINICAL TRIAL: NCT01698723
Title: A Double Blind Placebo Controlled Randomized Trial of Ribavirin in Patients With Acute on Chronic Liver Failure Due to Hepatitis E Virus
Brief Title: A Trial of Ribavirin in Patients With ACLF Due to Hepatitis E Virus
Acronym: HEVRibavirin
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Subrat Kumar Acharya, Professor, All India Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HEV-RIBA
Record Dates: First submitted 2012-09-27; First posted 2012-10-03 (Estimated); Last update posted 2016-04-26 (Estimated); Status verified 2016-04

CONDITIONS: Acute on Chronic Hepatic Failure; Liver Failure; Hepatitis E Infection
Keywords: ACLF; HEV; Ribavirin
MeSH Terms: conditions — Liver Failure | interventions — Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ribavirin (Active Comparator): 1000 mg (5 capsules)
  Interventions: Drug: Ribavirin
- Placebo (Placebo Comparator): 5 capsules of placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ribavirin
  Arms: Ribavirin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The term Acute on chronic liver failure (ACLF) describes a clinical entity characterized by an acute and rapid deterioration of liver function in a patient with previously well-compensated liver disease owing to the effects of a precipitating event. In this condition two insults act simultaneously, one being the preexisting liver injury (chronic liver disease) and the other acute injury which is responsible for the acute decompensation. HEV being a major factor responsible for this clinical entity and has a very high mortality rate. Ribavirin being a safe drug and has been shown to inhibit the replication of HEV, can be an important drug in the treatment of these patients. Therefore the present study is designed to study the impact of Ribavirin in reducing the mortality due to HEV related ACLF.

ELIGIBILITY:
Inclusion Criteria:

* All ACLF due to HEV
* Consent to participate in trial and collection of blood.

Exclusion Criteria:

* Pregnant and nursing mothers.
* Severe anemia
* Other etiologies of ACLF (eg. Alcohol, drugs, reactivation of hepatitis B and hepatitis C, variceal bleeding, surgical intervention and sepsis)
* Hepatocellular carcinoma (HCC)
* Hepatorenal syndrome (HRS) at admission
* Presence of life threatening cardiovascular, respiratory and neurological disease
* Acquired Immunodeficiency Syndrome
* Patients with hemoglobinopathies (e.g., thalassemia major, sickle-cell anemia)
* Refusal to provide consent to participate in the study

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Improvement in survival | 4 weeks and 12 moths

SECONDARY OUTCOMES:
Child Score | 4 weeks and 12 months
  Change in Child Score will be evaluated at every 4 week interval
Viremia | 4 weeks, 3 months
  Change in viral load
Variceal bleeding | 4 weeks and 12 months
  Variceal bleeding will be assessed every 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Subrat K Acharya, DM, Principal Investigator — All India Institute of Medical Sciences
Locations (2):
- India (2):
  - AII India Institute of Medical Sciences, Delhi, National Capital Territory of Delhi
  - All India Institute of Medical Sciences, Delhi, National Capital Territory of Delhi

IPD SHARING:
Plan to Share IPD: Yes